CLINICAL TRIAL: NCT05291988
Title: A Multilevel Approach to Improving Colorectal Cancer Screening in Rural Communities of the FH/UW Catchment Area
Brief Title: A Multilevel Approach for Improvement in Screening of Colorectal Cancer in Rural Communities, The Screen to Save Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RG1121686; NCI-2022-01172 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10786 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (S2S education, FIT kit) (Experimental): Participants receive S2S online screening education and FIT kit for sample collection.
  Interventions: Other: Educational Intervention; Other: Fecal Immunochemical Test; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive S2S education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Fecal Immunochemical Test — Receive FIT kit
  Other Names: FIT; iFOBT; immunoassay fecal occult blood test; immunochemical fecal occult blood test; Immunochemical FOBT; immunologic fecal occult blood test
Other: Questionnaire Administration — Ancillary Studies

SUMMARY:
This clinical trial determines the feasibility of a multilevel approach to improve colorectal cancer screening within two rural regions of the Fred Hutchinson Cancer Research Center/University of Washington Consortium catchment area. The catchment area is the greater Puget Sound Region (13 counties). These rural counties have the highest overall rates of cancer incidence and mortality in the area; rural/small town residents in the catchment area had the lowest rates of meeting mammogram, Pap, and colorectal screening recommendations. This study involves observational data and questionnaire assessments to determine if an online version of the evidence-informed national colorectal cancer screening program, known as "Screen to Save (S2S)" and a fecal immunochemical test (FIT) kit distribution are acceptable and accessible to patients. FIT kits may help doctors find colorectal cancer sooner, when it may be easier to treat.

DETAILED DESCRIPTION:
OUTLINE:

Participants receive S2S online screening education and FIT kit for sample collection.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years or older or < 45 years old with family history of CRC
* Speak and read English or Spanish
* Current resident in Clallam county
* Currently non-adherent to CRC screening recommendations

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Accessibility | Up to 3 months
  Three questions will be asked post-intervention to assess fit of the screen to save (S2S) education, suitability, and usefulness of the useful for learning about colorectal cancer (CRC) and CRC screening.
Acceptability | Up to 3 months
  Four questions will be asked post-intervention to assess approval, appeal, whether the participant liked, or welcomed the S2S education.
Participant uptake | Up to 3 months
  Feasibility evaluation will include assessment of the number of participants that respond to the letter of invitation to 1) participate in the educational portion of the project by viewing the online S2S education and completing the online questionnaires and 2) complete the pick-up and return of the FIT Kit. This will be assessed through participant tracking and follow-up procedures.
Demographic information | At pre-intervention only
  The following demographic information will be collected: participant's age, gender, race/ethnicity, preferred language, household income, highest level of education, insurance status, ZIP code, country of origin, and years of United States (U.S.) residence. Demographics will be analyzed within each group using Chi-square or Fisher's exact test for paired binary data.

SECONDARY OUTCOMES:
Colorectal cancer knowledge | Up to 3 months
  Knowledge will be assessed pre- and post-intervention. The knowledge scale will include 5 multiple choice knowledge questions about colorectal screening and colorectal cancer presented as part of the S2S inflatable colon education.
Behavioral intention | Up to 3 months
  Intention to get CRC screening will be assessed using one question with a 5-point response option (1 = Very Unlikely, 2 = Somewhat Unlikely, 3 = Neutral, 4 = Somewhat Likely, 5 = Very Likely).
Social engagement | Up to 3 months
  Social engagement likelihood will be measure using a single question about their intention to share information learned during the S2S education with others (parents, grandparents, relatives, peers, community members).
Medical and colorectal cancer information | At pre-intervention
  Use of regular health clinic and medical providers, history of colorectal cancer screening, and family and personal history of colorectal cancer diagnosis.
COVID-19 impact assessment | At pre-intervention
  A single question about the impact of COVID-19 on the decision to get colorectal cancer screening will determine if non-adherence was related to COVID-19. A yes/no response will be required.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ceballos, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT05291988/ICF_000.pdf